CLINICAL TRIAL: NCT04957680
Title: Effectiveness and Dissemination of Computer-based Cognitive Behavioral Therapy and Online Stress Management Program for Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBN2021
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- computer-based cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: CCBT
- online stress management program (Active Comparator)
  Interventions: Behavioral: CCBT
- waitlist (No Intervention)

INTERVENTIONS:
Behavioral: CCBT — computer-based treatment program for depressed adolescents
  Arms: computer-based cognitive behavioral therapy; online stress management program

SUMMARY:
The aim of this study is to investigate the effectiveness of a computer-based Cognitive Behavioral Therapy (CCBT) and online stress management program for adolescents, and identify the characteristics of depressed adolescents that participate in the programs.

ELIGIBILITY:
Inclusion Criteria:

* adolescents that scored above the threshold for mild depression (PHQ, CES-D)

Exclusion Criteria:

* adolescents with severe depression/neuropsychiatric conditions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
CES-D | 5 week
PHQ | 5 week

SECONDARY OUTCOMES:
DSM-5 Severity measure for Depression, Child-Adolescent version | 5 week
Perceived Stress Scale | 5 week
Study Stress Scale | 5 week
BAI | 5 week
EPQ | 5 week
Self-esteem Scale | 5 week
PedsQL 4.0 | 5 week
Homework compliance | 5 week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided